CLINICAL TRIAL: NCT05989529
Title: Uncovering Clinical Trial Engagement Among Individuals With Borderline Personality Disorder
Brief Title: Delving Into Borderline Personality Disorder Clinical Trial Experiences
Status: Not yet recruiting | Type: Observational
Sponsor: Power Life Sciences Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: 80910613
Record Dates: First submitted 2023-08-04; First posted 2023-08-14 (Actual); Last update posted 2023-08-14 (Actual); Status verified 2023-08

CONDITIONS: Borderline Personality Disorder
Keywords: borderline personality disorder
MeSH Terms: conditions — Borderline Personality Disorder

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Taking part in medical study usually favors a particular demographic group. But there is limited research available to explain what trial attributes affect the completion of these specific demographic groups.

This study will admit a wide range of data on the clinical research experience of borderline personality disorder patients to determine which factors prevail in limiting a patient's ability to join or finish a trial.

It will also try to analyze data from the perspective of different demographic groups to check for recurring trends which might yield insights for the sake of future borderline personality disorder patients.

ELIGIBILITY:
Inclusion Criteria:

* Aged ≥ 18 years old
* Clinical diagnosis of Borderline Personality Disorder
* Able to comprehend the investigational nature of the protocol and provide informed consent

Exclusion Criteria:

* No diagnosis of Borderline Personality Disorder confirmed
* Inability to perform regular electronic reporting
* Patient does not understand, sign, and return consent form

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with borderline personality disorder who are actively considering enrolling in an observational clinical trial but have not yet completed enrollment and randomization phases in said clinical trial.
Sampling Method: Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2024-09 (Estimated); Primary Completion 2025-09 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
Number of patients who decide to enroll in a borderline personality disorder clinical research | 3 months
Rate of patients who remain in borderline personality disorder clinical research to trial completion | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Michael B Gill, Study Director — Power Life Sciences Inc.
Locations (1):
- Power Life Sciences, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Garcia MC. [Treatment of borderline personality disorder with opioid antagonists: buprenorphine, nalmefene, naloxone and naltrexone in the treatment of dissociative symptoms, self-mutilation and suicidal behavior]. Vertex. 2020 Apr;XXX(148):1-10. doi: 10.53680/vertex.v30i148.122. Spanish. PMID 33890928
- [Background] Kvarstein EH, Froyhaug M, Pettersen MS, Carlsen S, Ekberg A, Fjermestad-Noll J, Ulvestad DA, Gikling EL, Hjermann E, Lindberget K, Omvik S, Eikenaes IU, Hummelen B, Morken KTE, Wilberg T, Pedersen GAF. Improvement of personality functioning among people treated within personality disorder mental health services. A longitudinal, observational study. Front Psychiatry. 2023 May 9;14:1163347. doi: 10.3389/fpsyt.2023.1163347. eCollection 2023. PMID 37229394
- [Background] Jacob GA, Hauer A, Kohne S, Assmann N, Schaich A, Schweiger U, Fassbinder E. A Schema Therapy-Based eHealth Program for Patients with Borderline Personality Disorder (priovi): Naturalistic Single-Arm Observational Study. JMIR Ment Health. 2018 Dec 17;5(4):e10983. doi: 10.2196/10983. PMID 30559092

DOCUMENTS (1):
  • Informed Consent Form (2023-08-04): https://cdn.clinicaltrials.gov/large-docs/29/NCT05989529/ICF_000.pdf